CLINICAL TRIAL: NCT00447434
Title: An Open-Label, Parallel Comparison Study to Evaluate the Effect of Oral Administration of Nattokinase Taken by Normal Subjects, Patients Under Dialysis, and Patients of Cardiovascular High Risk Groups
Brief Title: Efficacy and Safety of Natto Extract
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I050308
Record Dates: First submitted 2007-03-13; First posted 2007-03-14 (Estimated); Last update posted 2007-03-14 (Estimated); Status verified 2007-03

CONDITIONS: Thrombosis; Cardiovascular Diseases
Keywords: Nattokinase; fibrinolytic factors; blood lipids; nutrimental supplement
MeSH Terms: conditions — Thrombosis; Cardiovascular Diseases | interventions — Soy Foods; nattokinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Natto extract (Nattokinase)

SUMMARY:
Nattokinase is a potent fibrinolytic enzyme extracted from Natto. The objective of this study was to compare the efficacy of the natto extract taken by healthy volunteers, dialysis patients, and patients with cardiovascularrisk factors on the fibrinolytic factors and blood lipids. The study has two primary objectives: to evaluate the effect of oral intake of nattokinase in normal subjects, patients under dialysis, and patients of cardiovascular high risk group, and to compare the effect of oral intake of nattokinase among three groups.

Fifteen subjects, 20-70 years, for each group will be enrolled to take the capsules of natto extract orally for 2 months. Fibrinolytic factors, vital signs and blood lipids for efficacy, and body weight, renal function and self-administered questionnaire for safety will be assessed at screening, 3, 7, 28, and 56 days after the initiation of intake, and 2 weeks after the cease of intake.

DETAILED DESCRIPTION:
This study will employ an open-label, parallel-group design. Adult men and women who meet the inclusion/exclusion criteria and give written consent to participate will be assigned to one of the three groups according to their condition: Group A- normal volunteers; Group B- patients under dialysis; Group C- patients of cardiovascular high risk group. Each group will enroll 15 subjects. After two to four weeks run-in period, subjects will be given nattokinase orally for 8 weeks, and will be asked to stop taking nattokinase for 2 weeks to evaluate the effect of long-term intake and cease of intake of nattokinase.

Laboratory tests, including fibrinogen, T-PA, PAI-1, D-dimer, total cholesterol, LDL-C, HDL-C, and TG, vital signs and body weight will be evaluated at screening visit, 3 days, 1 week, 4 weeks, 8 weeks, and 10 weeks (2 weeks after cease of intake) visits. Patient self-evaluation of tolerance and physical improvement will be assessed by a Patient Questionnaire at 3-day, and 1-, 4-, 8-, and 10-week visits. Each patient will be carefully monitored for the development of any adverse events (AE).

ELIGIBILITY:
Inclusion Criteria:

* In order to be enrolled in the study, potential study subjects must meet the following inclusion criteria:

  1. Men and non-pregnant women who are at least 20 and younger than 70 years of age.
  2. Subjects who are, in the opinion of the Investigator, able to comply with the requirements of the study.
  3. Subjects who have been adequately informed of the nature and risks of the study and who have given written informed consent prior to receiving investigational product.

Group-specific inclusions criteria:

Group A:

1. Subjects have no risk factors of cardiovascular diseases (see Group C) or chronic renal diseases in the history.
2. Male subjects have Creatinine≦1.4 mg/dl; Female≦1.3 mg/dl.

Group B:

1. Patients have been receiving dialysis at the same institute for at least 3 months.

Group C:

1. Patients have coronary artery disease (CAD); OR
2. Patients have peripheral arterial occlusive disease (PAOD); OR
3. Patients have history of stroke; OR
4. Patients have history of transient ischemic attack (TIA); OR
5. Patients have history of pulmonary embolism (PE); OR
6. Patients have history of deep vein thrombosis (DVP); OR
7. Patients have more than 2 major risk factors of cardiovascular disease (CVD) listed by National Health Insurance guidelines such as hypertension, smoking, diabetes mellitus (DM), atrial fibrillation (AF), lipid disorder, overweight, physical inactivity, etc.

Exclusion Criteria:

* In order to be enrolled in the study, potential study patients must not have any of the following exclusion criteria:

  1. Known allergies to the component of study product.
  2. Current use of warfarin.
  3. Patients have active disease status.
  4. Patients have acute disease, and in the opinion of investigators, are not suitable to participate in this study.

Group-specific exclusion criteria:

Group A:

1. Patients have coronary artery disease (CAD).
2. Patients have peripheral arterial occlusive disease (PAOD).
3. Patients have history of stroke.
4. Patients have history of transient ischemic attack (TIA).
5. Patients have history of pulmonary embolism (PE).
6. Patients have history of deep vein thrombosis (DVP).
7. Patients have more than 2 major risk factors of cardiovascular disease (CVD) listed by National Health Insurance guidelines such as hypertension, smoking, diabetes mellitus (DM), atrial fibrillation (AF), lipid disorder, overweight, physical inactivity, etc.
8. Patients have history of chronic renal diseases.
9. Male subjects have Creatinine>1.4 mg/dl; Female>1.3 mg/dl.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-06; Study Completion 2005-10

PRIMARY OUTCOMES:
fibrinolytic factors
vital signs
blood lipids

SECONDARY OUTCOMES:
renal function
body weight
self-administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsun Hsia, MD, Principal Investigator — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan